CLINICAL TRIAL: NCT06125990
Title: Effect of Video Game-Based Lung Volume Increasing Training on Respiratory Mechanics in Children With Developmental Delays: Randomized Controlled Study
Brief Title: Video Based Breathing Exercise Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VideoBasedRehab
Record Dates: First submitted 2023-09-18; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder; Down Syndrome
Keywords: breathing exercise; video based game; biofeedback
MeSH Terms: conditions — Autism Spectrum Disorder; Down Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Each children were be interviewed and evaluated alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (SGr) (Experimental): In addition to institutional conventional rehabilitation, this group included breathing exercises to increase lung volumes and a 21-minute breathing exercise with video-based biofeedback.
  Interventions: Other: Experimental: Study Group (SGr)
- Control Group (CGr) (Sham Comparator): This group was given only institutional conventional rehabilitation.
  Interventions: Other: Sham Comparator: Control Group (CGr)

INTERVENTIONS:
Other: Experimental: Study Group (SGr) — For 6 weeks, in addition to institutional conventional exercise 2 days a week, one day a week of home exercise, breathing exercises to increase lung volumes and 7 sets of video-based breathing exercises were applied, each set consisting of 2 minutes of performance and 1 minute of rest.
  Arms: Study Group (SGr)
Other: Sham Comparator: Control Group (CGr) — Only institutional conventional rehabilitation was implemented.
  Arms: Control Group (CGr)

SUMMARY:
The aim of the study was to investigate the effect of video game-based lung volume increasing training on respiratory mechanics in children with developmental delays. Individuals with special needs are people who, for various reasons, show significant awareness at the level expected from their peers in terms of their individual characteristics and educational qualifications. Individuals with special needs constitute an important part of our country. Children with special needs may have respiratory problems that may or may not be recognized because they are not diagnosed, as well as decreases in respiratory capacity. Decrease in lung volumes may be encountered in children with special needs with various diagnoses such as neuromuscular diseases, cerebral palsy, cystic fibrosis, autism, and Down syndrome.

Pulmonary rehabilitation is a multidisciplinary program that balances or reverses the physiopsychopathology of pulmonary disorders and tries to help the patient reach high functional capacity as much as his physical condition and pulmonary disability allow. Chest physiotherapy, which is an important step of pulmonary rehabilitation, is a rehabilitation intervention used to reduce airway resistance, improve gas exchange and facilitate breathing in children. Active video game systems produced with the development of new technologies are used for the positive progression of rehabilitation, especially in young individuals who are extensive users of digital devices. For children who need a pulmonary rehabilitation program, active video game systems are preferred in the clinic as they increase the compatibility of the sessions and ensure continuity.

DETAILED DESCRIPTION:
It seems that there are insufficient studies in the literature on the effects of exercises that increase lung capacity on children with special needs. To the best of our knowledge, there is no study investigating the effects of programs to increase lung volumes in children with special needs in a randomized controlled study design. With this project, we aimed to reveal the effects of a lung volume-increasing exercise program performed with a video-based game system applied for 6 weeks in children with special needs, by comparing it with the control group that received only conventional rehabilitation. The duration of the treatment program in our study is also one of our unique values. According to our literature research, the implementation of a lung capacity-increasing rehabilitation program in children with special needs in the form of supervision twice a week and a home program once a week for 6 weeks is the first.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer of the family to participate in the study
* Stable clinical status at inclusion without infection or exacerbation in the previous 4 weeks
* Children who have not been included in another clinical trial within the last month
* Participants with a Body Mass Index (BMI) below 30 kilograms/square meter

Exclusion Criteria:

* Those with severe comorbidities, unstable coronary artery disease, collagen vascular diseases, and those requiring high-flow oxygen therapy (3-4 L\min).
* History of exertional syncope or any comorbidity that prevents exercise training
* Inability to communicate with the child and the child not obeying commands in any way
* Children with vision problems

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
FVC Measurement | Change from baseline lungs volumes at 6 weeks.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.
FEV1 Measurement | Change from baseline lungs volumes at 6 weeks.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.
FEV1/FVC Measurement | Change from baseline lungs volumes at 6 weeks.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.
PEF Measurement | Change from baseline lungs volumes at 6 weeks.
  Respiratory Function Test. The COSMED microQuark spirometer used. Positive airway flow rate was evaluated.

SECONDARY OUTCOMES:
Pulse measurement | Change from baseline lungs volumes at 6 weeks.
  In order to ensure exercise safety, exercise sessions were carried out by monitoring pulse and saturation values with a pulse oximeter before, during and during exercises that increase lung volumes.
Saturation measurement | Change from baseline lungs volumes at 6 weeks.
  In order to ensure exercise safety, exercise sessions were carried out by monitoring pulse and saturation values with a pulse oximeter before, during and during exercises that increase lung volumes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gedik University Barrier-Free Life Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simmich J, Deacon AJ, Russell TG. Active Video Games for Rehabilitation in Respiratory Conditions: Systematic Review and Meta-Analysis. JMIR Serious Games. 2019 Feb 25;7(1):e10116. doi: 10.2196/10116. PMID 30801256
- [Background] Ucgun H, Gurses HN, Kaya M, Cakir E. Video game-based exercise in children and adolescents with non-cystic fibrosis bronchiectasis: A randomized comparative study of aerobic and breathing exercises. Pediatr Pulmonol. 2022 Sep;57(9):2207-2217. doi: 10.1002/ppul.26026. Epub 2022 Jun 21. PMID 35669989